CLINICAL TRIAL: NCT00074360
Title: The Effect of Ethanol on Cerebral Blood Flow as Measured by Functional Magnetic Resonance Imaging and the Development of Conditioned Response to Ethanol Administration
Brief Title: The Effect of Ethanol on Brain Activity
Status: Completed | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040060; 04-AA-0060
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2012-12-17

CONDITIONS: Healthy
Keywords: Ethanol; fMRI; Blood Flow; Conditioning; Reinforcement

SUMMARY:
This study is divided into two parts; each designed to answer a separate but related question:

Which brain regions are activated in humans by the rewarding properties of ethanol administration?

Is it possible to demonstrate a conditioned response to a stimulus paired with rising blood alcohol concentrations (BAC) in humans and can this response be observed in the brain using functional magnetic resonance images (fMRI) techniques?

Part 1. In order to determine which brain regions are activated by the rewarding properties of ethanol administration, we propose to use Blood Oxygenation Level Dependent (BOLD) fMRI techniques to test the hypothesis that during the time of rising and peak BAC, mesolimbic, mesocortical, and nigrostriatal dopamine (DA) terminal areas of the brain will show significant increases in cerebral blood flow. Healthy, non-alcoholic subjects will be given intravenous (IV) ethanol or placebo infusions on separate days. The infusions will have three phases. On each day, during the first phase a saline infusion will be used to measure basal brain blood flow. The second phase will be an ethanol infusion delivered at rates calculated to produce a BAC of 0.08 plus or minus 0.005 g/dl at 10 minutes. The rate of the infusion for the next 10 minutes (third phase) will be calculated to maintain BAC at the target level of 0.08 plus or minus 0.005 g/dl for the duration of the infusion. On the placebo day, subjects will receive a saline infusion at the same set of rates for phases two and three as used during their ethanol infusion. Continuous multi-slice fMRI data will be collected during each infusion.

Part 2. In order to investigate conditioned response to ethanol, three groups of healthy, non-alcoholic subjects will be given a series of IV infusions on separate days. The experimental group will receive ethanol infusion paired with a conditioned stimulus (CS) which will be presented while the BAC is rising. One control group (I) of healthy, non-alcoholic subjects will also be given a series of intravenous ethanol infusions on separate days, but these infusions will not be paired with a CS. The other control group (II) will be given only saline infusions during the CS presentation. After three training sessions, all three groups will undergo an fMRI scan during which the CS will be paired with saline infusion. This will allow the response to the CS alone to be observed. After 10 minutes of CS presentation, the ethanol infusion will begin and continue for another 15 minutes. Conditioned response (CR) will be demonstrated if the experimental group shows greater increase in BOLD signal than the control groups in motivation areas such as mesolimbic, mesocortical, and nigrostriatal dopamine (DA) terminal areas of the brain in response to the CS while they receive the saline infusion. Control group II will also undergo an fMRI scan and will be given saline infusion followed by ethanol infusion during their last 15 minutes in the scanner to control for the non-specific effects of repeated infusions & scans on BOLD response to ethanol. If we are able to produce a CR in brain regions associated with motivation, it may be possible to use this CR as an experimental model for human alcohol craving.

DETAILED DESCRIPTION:
This study is designed to answer four questions:

1. Which brain regions are activated in humans by the rewarding properties of ethanol administration?
2. How does ethanol administration affect the brain response to visual cues known to evoke positive or negative emotion?
3. Do individuals who regularly drink in ethanol in large amounts (heavy drinkers) differ from individuals who do not regularly drink large amounts of ethanol (social drinkers) in how ethanol affects brain function?
4. Does ethanol administration affect the brain regions activated in a risk-taking task in social drinkers and heavy drinkers?

In order to determine which brain regions are activated by the rewarding properties of ethanol administration, we propose to use Blood Oxygenation Level Dependent (BOLD) fMRI techniques to test the hypothesis that during the time of rising and peak BAC, mesolimbic, mesocortical, and nigrostriatal dopamine (DA) terminal areas of the brain will show significant increases in cerebral blood flow. Healthy, subjects who are not seeking treatment for an alcohol use disorder will be given intravenous (IV) ethanol or placebo infusions on separate days. An ethanol infusion will delivered at rates calculated to produce a BAC of 0.08 plus or minus. An ethanol infusion will delivered at rates calculated to produce a BAC of 0.08 plus or minus 0.005 g/dl at 15 minutes. Then the rate of the infusion will be adjusted so that for the next 30 minutes (second phase) BAC will be maintained at the target level of 0.08 0.005 g/dl. On the placebo day, subjects will receive a saline infusion at the same set of rates as used during their ethanol infusion. Continuous multi-slice fMRI data will be collected during each infusion. During each infusion, BOLD response to visual stimuli designed to evoke emotion will also be examined. In addition, we will compare the BOLD response of healthy social drinkers to that of healthy heavy drinkers. We will also compare the BOLD response elicited by risk-taking during the ethanol infusion to that during the placebo infusion in both social and heavy drinkers.

ELIGIBILITY:
* INCLUSION CRITERIA LIGHT DRINKERS:

  1. in good health.
  2. between 21 and 45 years of age.

     <TAB>
  3. Currently consuming between 1 and 14 drinks per week.

EXCLUSION CRITERIA LIGHT DRINKERS:

1. have an abnormal physical exam and/or have laboratory values outside of normal ranges;
2. have fulfilled DSM-IV criteria for ethanol or other substance dependency (excluding nicotine) at any time;
3. have fulfilled DSM-IV criteria for a current or past major psychiatric disorder (DSM-IV Axis I) or who have ever had a head injury requiring hospitalization.
4. are over or under 20% of ideal body weight;
5. have taken any prescribed, non-prescribed, or over-the-counter medications or drugs within 14 days prior to the study days (excluding oral contraceptive agents);
6. are pregnant;
7. report to have a "facial flushing" response to the consumption of ethanol;
8. have never consumed at least two standard drinks of ethanol within one hour.
9. have ferromagnetic objects in their bodies, which might be adversely affected by MRI (e.g., surgical clips, metal fragments in or near brain, eye or blood vessels, cardiac or neurological pacemaker, cochlear or eye implant). Any doubt about presence of these objects will result in exclusion from this study.
10. Additionally, subjects will be asked to abstain from ethanol for at least 2 days prior to the studies.
11. Regular tobacco users will be excluded from the study in order to avoid nicotine withdrawal symptoms. Occasional (not daily) use of tobacco products is acceptable.

INCLUSION CRITERIA HEAVY DRINKERS:

1. in good health.
2. between 21 and 45 years of age.
3. currently consuming between 20 and 40 drinks per week.
4. not regularly abstinent for more than 3 days per week, but have abstained from alcohol for 3 consecutive days without experiencing withdrawal symptoms.
5. able to provide a plausible history that they can abstain from alcohol without significant withdrawal symptoms when coming to the clinic. In addition, each participant will be asked to quantify their worst withdrawal symptoms using the Clinical Institute Withdrawal Assessment (CIWA) Instrument. Participants who score 8 or above will not be enrolled in the protocol.
6. not seeking treatment for their alcohol consumption.

EXCLUSION CRITERIA HEAVY DRINKERS:

1. have an abnormal physical exam and/or have laboratory values outside of normal ranges;
2. have fulfilled DSM-IV criteria for any substance dependency (excluding alcohol or nicotine) at any time;
3. have fulfilled DSM-IV criteria for a current or past major psychiatric disorder or who have ever had a head injury requiring hospitalization.
4. are over or under 20% of ideal body weight;
5. have taken any prescribed, non-prescribed, or over-the-counter medications or drugs within 14 days prior to the study days (excluding oral contraceptive agents);
6. are pregnant;
7. report to have a "facial flushing" response to the consumption of ethanol;
8. have never consumed at least two standard drinks of ethanol within one hour.
9. have ferromagnetic objects in their bodies, which might be adversely affected by MRI (e.g., surgical clips, metal fragments in or near brain, eye or blood vessels, cardiac or neurological pacemaker, cochlear or eye implant). Any doubt about presence of these objects will result in exclusion from this study.
10. Additionally, subjects will be asked to abstain from ethanol for at least 2 days prior to the studies.
11. Regular tobacco users will be excluded from the study in order to avoid nicotine withdrawal symptoms. Occasional (not daily) use of tobacco products is acceptable.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2003-12-09; Study Completion 2012-12-17

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Hommer, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Blekher T, Ramchandani VA, Flury L, Foroud T, Kareken D, Yee RD, Li TK, O'Connor S. Saccadic eye movements are associated with a family history of alcoholism at baseline and after exposure to alcohol. Alcohol Clin Exp Res. 2002 Oct;26(10):1568-73. doi: 10.1097/01.ALC.0000033121.05006.EF. PMID 12394291
- [Background] Boileau I, Assaad JM, Pihl RO, Benkelfat C, Leyton M, Diksic M, Tremblay RE, Dagher A. Alcohol promotes dopamine release in the human nucleus accumbens. Synapse. 2003 Sep 15;49(4):226-31. doi: 10.1002/syn.10226. PMID 12827641
- [Background] Breiter HC, Gollub RL, Weisskoff RM, Kennedy DN, Makris N, Berke JD, Goodman JM, Kantor HL, Gastfriend DR, Riorden JP, Mathew RT, Rosen BR, Hyman SE. Acute effects of cocaine on human brain activity and emotion. Neuron. 1997 Sep;19(3):591-611. doi: 10.1016/s0896-6273(00)80374-8. PMID 9331351